CLINICAL TRIAL: NCT00361907
Title: Effect of Pulsatile IV Insulin Delivery on Circulating Risk Markers of Vascular and Metabolic Complications in Pts With Diabetes
Brief Title: Effect of Pulsatile IV Insulin on Circulating Risk Markers of Vascular and Metabolic Complications in Pts With Diabetes
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Administrative - Suspended by IRB
Sponsor: Florida Atlantic University (Other)
Collaborators: Advanced Diabetes Treatment Centers (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H09-04; MH42900 and MH01386 (Other: NIMH)
Record Dates: First submitted 2006-04-13; First posted 2006-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus
Keywords: Pulsatile intravenous insulin; Oral carbohydrate loading; Respiratory Quotients; Hypoglycemia; Diabetic Complications; Circulating vascular and inflammatory markers
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Diabetes Complications | interventions — Insulin, Regular, Human; Insulin Aspart

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Diabetic patients who meet inclusion criteria will be enrolled to start Pulsatile Intravenous Insulin Therapy on a weekly basis. Baseline testing will be performed and measured against continued testing every twelve months.
  Interventions: Procedure: Effect of Pulsatile IV insulin on diabetic pt blood markers
- 1 (Placebo Comparator): Circulating blood markers will be performed on diabetic control patients at baseline and every twelve months to compare and measure against patients treated with Pulsatile intravenous insulin therapy
  Interventions: Procedure: Effect of Pulsatile IV Insulin on blood markers; Procedure: Effect of Pulsatile IV insulin on diabetic pt blood markers

INTERVENTIONS:
Procedure: Effect of Pulsatile IV insulin on diabetic pt blood markers — Diabetic patients are given pulsatile intravenous insulin on a weekly basis determined by weekly physician order based on pt response and insulin resistance.
  Other Names: Humulin, Humulog, Novolog, Epidra
  Arms: 2
Procedure: Effect of Pulsatile IV Insulin on blood markers — Circulating blood markers are performed at baseline and every twelve months to compare and measure against diabetic patients receiving pulsatile intravenous insulin.
  Arms: 1
Procedure: Effect of Pulsatile IV insulin on diabetic pt blood markers — Blood markers will be performed on diabetic patients enrolled as control patients at baseline and every twelve months to measure and compare against diabetic patients treated with Pulsatile intravenous insulin therapy
  Arms: 1

SUMMARY:
The purpose of this study is to determine the effect of Pulsatile Intravenous Insulin therapy on circulating blood markers. These blood markers are selected due to their correlation to and possible pathogenetic roles in vascular compromise and inflammatory malfunction in diabetic patients.

DETAILED DESCRIPTION:
Insulin produces vasodilatory, anti inflammatory and anti thrombotic effects (1-4). . However the effects of pulsatile intravenous insulin delivery on circulating risk factors for vascular and metabolic disease is unknown. This study is used to evaluate circulating risk markers of vascular and metabolic disease compared to a matched control group.

Protocol Patients selected have diabetes mellitus, 20 years of age and older, and are treated with oral agents and/or insulin. The study is for a minimum of 12 months and may continue for 2-3 years if a significant difference is shown following the initial 12 months. Blood markers will be determined every 12 months for the first year, and every 12 months after that. They may include the following: BNP, fructosamine, PAI-1, fibrinogen, homocysteine, endothelin 1, aldosterone, VCAM, ICAM, IGF-1, TGF-beta, TNF-alpha, hs-CRP, and IL-6). The results are compared to an age and fructosamine matched control group.

Endpoints; Changes in markers Statistics: ANOVA Blood: 2 purple, 2 red, 2 blue tops

The respiratory quotient (RQ) is a measurement of CO2 exhaled and O2 inhaled and is proportionate to the fuel sources being used by the body, primarily the liver over short periods of time. The higher the RQ, the more glucose and less alternative fuel sources are being utilized. Following the RQ change helps determine the effectiveness of physiological insulin administration in increasing anabolic functions in diabetic individuals. By improving the body's glucose metabolism and thereby causing beneficial effects of anabolic factors, the possibility of serious complications can be decreased. In addition the use of oral carbohydrate at the same time along with the physiologic insulin administration stimulates the appropriate gut hormones which augment this effect, a response which cannot be duplicated with intravenous glucose. The purpose of our studies is to determine whether the physiologic administration of pulsatile intravenous insulin along with the augmenting effect of oral carbohydrates will normalize metabolism in diabetic patients and improve their quality of life indices.

The RQ is determined by the use of a metabolic cart. Individuals breathe into a mask for 3-5 minutes after a rest period of 30 or more minutes. The ratio of exhaled volume of CO2 to the inhaled volume of O2 is determined as the RQ. The physiologic range is 0.7 to1.3. Individuals using fat as a primary fuel have a ratio of 0.7, protein or mixed fuels is 0.8-0.9 and carbohydrate is 0.9-1.0. Those taking excessive calories will have RQ's higher than 1.05. The RQ can be followed serially and this is done twice, before and after each treatment, during the 3 successive sessions on a single treatment day. The amount of intravenous insulin and oral glucose given is determined by the RQ changes during the previous session.

Pusatile intravenous insulin delivery is a process which encourages the glucose metabolism in diabetics to normalize in multiple organs, especially muscle, retina, liver, kidney and nerve endings. The process fundamentally requires the administration of high dose intravenous insulin pulses similar to those found in non diabetic humans by their pancreas into the surrounding portal circulation. Oral carbohydrates are given simultaneously to augment the process and prevent hypoglycemia. The process is monitored by frequent glucose level measurements and respiratory quotients (RQ). RQ is measured by a metabolic cart which determines the ratio VCO2/ VO2. This ratio is specific for the fuel used at any one time by the body. The glucose levels are monitored to keep glucose levels appropriate and the RQ determines the need to readjust the infusion protocol in each patient for subsequent insulin infusion sessions. Pulsatile intravenous insulin delivery is done over 1-hour periods with a up to a 1-hour rest period between each session for three courses each day of activation.

References:

Katakam PVG, Tulbert CD, Snipes JA, Erdos B, Miller AW, Busija DW, Impaired Insulin-induced Vasodilation in Small Coronary Arteries of Zucker Obese rats is Mediated by Reactive Oxygen Species, AJP-Heart 288:854-60, 2005.

Chakraborty K Sinha AK, The Role of Insulin as an Antithrombotic Humoral Factor, BioEssays 26:91-98, 2003.

Elias AN, Eng S, Homocysteine Concentrations in Patients with Diabetes Mellitus-Relationship to Microvascular and Macrovascular Disease, Diabetes, Obesity and Metabolism 7:117-21, 2005.

Patiag D, Qu X, Gray S, Idris I, Wilkes M, Seale JP, Donnely R, Possible Interactions between Angiotensin II and Insulin:Effects on Glucose and Lipid Metabolism in vivi and in vitro, Journal of Endocrinology 167: 525-31, 2000

ELIGIBILITY:
Inclusion Criteria:

* We will include up to 500 patients both male and female over the age of 21 diagnosed with type 1 or type 2 diabetes mellitus
* All patients must have secondary complications caused by the diabetes and not responding to conventional medical management
* Under an Endocrinologists supervision for their diabetes management
* Endocrinologist must assess and approve patient for participation in this study
* Ability to swallow without difficulty
* Ability to commit to the weekly time requirements associated with the study

Exclusion Criteria:

* Other causes of complications not related to diabetes
* Lack of intravenous access
* Pregnancy
* Alcohol abuse, drug addiction or the use of illegal drugs
* Positive HIV
* Inability to perform breathe into machine for respiratory quotients

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2005-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Primary: Assessment of effect of Pulsatile Intravenous Insulin therapy on circulating blood markers for diabetic patients. | Circulating blood markers will be drawn at baseline and every twelve months to monitor and measure results

CONTACTS AND LOCATIONS:
Overall Officials: Betty Tuller, Ph.D, Principal Investigator — Florida Atlantic University
Locations (1):
- Florida Atlantic University Center for Complex Systems and Brain Sciences, Boca Raton, Florida, United States

REFERENCES:
- [Background] Hanke CJ, Drewett JG, Myers CR, Campbell WB. Nitric oxide inhibits aldosterone synthesis by a guanylyl cyclase-independent effect. Endocrinology. 1998 Oct;139(10):4053-60. doi: 10.1210/endo.139.10.6252. PMID 9751482
- [Background] Mather KJ, Lteif A, Steinberg HO, Baron AD. Interactions between endothelin and nitric oxide in the regulation of vascular tone in obesity and diabetes. Diabetes. 2004 Aug;53(8):2060-6. doi: 10.2337/diabetes.53.8.2060. PMID 15277386
- [Background] Ellis G, Adatia I, Yazdanpanah M, Makela SK. Nitrite and nitrate analyses: a clinical biochemistry perspective. Clin Biochem. 1998 Jun;31(4):195-220. doi: 10.1016/s0009-9120(98)00015-0. PMID 9646943